CLINICAL TRIAL: NCT02886247
Title: National Familial Pancreas Tumor Registry
Brief Title: Pancreatic Cancer Registry: For Any Person With a Personal or Family History
Acronym: NFPTR
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NA_00035453; P50CA062924 (NIH)
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Pancreatic Cancer, ATM, BRCA, Hereditary Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Hereditary Sensory and Autonomic Neuropathies

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and saliva
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- participants: individuals with a personal or family history of pancreas tumors

SUMMARY:
The NFPTR was established in 1994 to find the causes of pancreatic cancer. In brief, the investigators are interested in both the genetic and non-genetic causes of pancreatic cancer. The investigators are particularly interested in finding the genes that cause pancreatic cancer to cluster in some families. Up to 10% of pancreatic cancer patients have another close relative who has also developed pancreatic cancer. This clustering of pancreatic cancers in families has yet to be explained; however, the investigators continue to identify new familial pancreatic cancer genes that explain this clustering in subsets of families. For example, in 2009 and 2012 the investigators discovered that mutations in the PALB2 and ATM genes jointly account up to 5% of the clustering of pancreatic cancer in families.

ELIGIBILITY:
Inclusion Criteria:

* personal or family history of pancreas tumors

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: individuals with a personal or family history of pancreas tumors
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 1994-06; Primary Completion 2030-06 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
pancreatic cancer | 35 years

CONTACTS AND LOCATIONS:
Overall Officials: Alison Klein, PhD, MHS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States